CLINICAL TRIAL: NCT00042692
Title: Catechol Thioethers in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 10196-CP-001
Record Dates: First submitted 2002-08-05; First posted 2002-08-06 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Parkinson's Disease
Keywords: catechol thioethers; Parkinson's disease; neurodegenerative disease
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The goal of the clinical trial aim in this project is to test whether catechol thioethers can be used as biomarkers of dopaminergic neurodegeneration.

ELIGIBILITY:
First diagnosis of Parkinson's disease.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2001-03; Study Completion 2002-03